CLINICAL TRIAL: NCT02463695
Title: Characterisation of Cortical Vestibular Evoked Potentials (C-VEPs): A Comparative Study of Normal Ears Versus Those With Vestibular Deficits
Brief Title: Characterisation of Cortical Vestibular Evoked Potentials (C-VEPs)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STH18541
Record Dates: First submitted 2015-05-28; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Vestibular Neuronitis
Keywords: partial vestibular deficit; cortical vestibular evoked potential
MeSH Terms: conditions — Vestibular Neuronitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- vestibular deficit (Experimental): * Initial clinical assessment including otoneurological examination, pure tone audiometry, tympanometry vestibular screening tests and Magnetic Resonance Imaging as clinically indicated.
  * The cortical vestibular evoked potentials will add approximately add an extra 30 minutes to the test sequence but is minimally invasive and will not cause any pain or discomfort. It will be conducted on both the affected and non-affected ears.
  Interventions: Procedure: cortical vestibular evoked potentials (CVEPs)
- otologically normal controll (Active Comparator): Normative data will be collected from 36 normal ears from subjects that have no history of audiovestibular symptoms and are not being investigated for any balance disorders. The cortical vestibular evoked potentials will be recorded from both ears
  Interventions: Procedure: cortical vestibular evoked potentials (CVEPs)

INTERVENTIONS:
Procedure: cortical vestibular evoked potentials (CVEPs) — CVEPs utilise an existing method used to interrogate cortical projections from the auditory system in which sound waves stimulate the inner ear and the resulting electrical responses from the brain are recorded (known as Cortical Auditory Evoked Potentials CAEPs)
  Other Names: Cortical auditory evoked potential

SUMMARY:
The pathophysiology of vertigo is complex and usually requires specialist involvement. During the diagnostic process, patients commonly undergo tests which assess the integrity of the gaze and posture stabilisation mechanisms involving the inner ear (vestibular system), the visual systems and the subconscious neural pathways that interconnect them. Whilst these tests are useful they fail to provide information concerning the neural connections to the cortex and therefore neglect the perceptual aspects of disequilibrium.

At present the possibility of routine examination of these higher projections remains elusive as no practical alternatives to the expensive functional magnetic resonance imaging systems exist. However, recently a novel method of recording cortical vestibular evoked potentials (CVEPs) has been described.

CVEPs utilise an existing method used to interrogate cortical projections from the auditory system in which sound waves stimulate the inner ear and the resulting electrical responses from the brain are recorded. The recent breakthrough is in the realisation that these responses also contain information from the balance organs and therefore are a direct measure of cortical processing of the vestibular inputs.

Current evidence shows that CVEPs are present in the normal population and absent in patients with no vestibular function. The primary aim for this study is to extend the patient cohort to include those who have a vestibular injury but retain residual function. Patients going through standard testing will have also have CVEPs on both ears providing seminal information into the effect of injury to the peripheral vestibular system on the cortical pathways. Furthermore, by following the cohort through their complete management pathway it will be possible to ascertain if the CVEP can be used to predict rehabilitation outcome success.

DETAILED DESCRIPTION:
Ears with a vestibular deficit:

Patients referred to the tertiary ear nose and throat clinics as well otoneurological clinics at the Royal Hallamshire will be eligible for enrolment. The investigators aim to record data from 36 ears with vestibular dysfunction.

A) Patients will receive a consultation with an ENT Consultant or Registrar as per standard practice.

B) If the patient is deemed by the doctor to have an otoneurological cause for their symptoms then further audiovestibular testing and imaging will be arranged as per standard practice. The patients will then be made aware of this study and if interested will be given the opportunity to discuss it further with the chief investigator (CI) or the principal investigator (PI).

C) If agreeable the patients will be given information packs by the PI/CI and taken through the study.

D) The patients will leave the consultation with the information pack and be asked to consider participation in the study. They will have no obligation to take part and they can contact the any member of the research team to ask for further information or to have any questions answered.

E) Upon their return for audiovestibular testing the patients will inform the CI/PI if they wish to participate in the study and if so will have an additional test at the end of test sequence. This will add approximately 30 minutes to their appointment time.

F) Patients who are suitable for rehabilitation (as per standard care pathway) will go ahead and have the course of treatment at subsequent visit(s). The outcomes following the treatment will be logged and correlated with the CVEP to check for any correlation that may or may not be present.

Otologically normal ears:

Normative data will be collected from 36 normal ears from subjects that have no history of audiovestibular symptoms and are not being investigated for any balance disorders. Healthy controls will be recruited via poster advertisements and potential participants asked to contact the research team if they are considering taking part.

ELIGIBILITY:
Inclusion Criteria:

* Vestibular deficit Group:

  1. Over 18 years of age
  2. Can provide informed consent
  3. Deemed to have an otoneurological cause for their symptoms (true vertigo, room spinning even when head is still)
  4. No middle ear pathology

NORMATIVE GROUP:

1. Over 18 years of age
2. Can provide informed consent
3. No previous otoneurological history

Exclusion Criteria:

* VESTIBULAR DEFICIT GROUP PATIENTS

  1. Participants under the age of 18
  2. Participants unable to provide informed consent
  3. Patients not deemed to have an otoneurological cause for their symptoms
  4. Patients with middle ear pathology

NORMATIVE GROUP:

1. Previous history of problems with hearing and or balance
2. Participants under the age of 18
3. Participants unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The degree of change of cortical vestibular evoked potential measured by amplitude (in microvolts) | 6 months

SECONDARY OUTCOMES:
The time interval between the stimulation and response (latency) of cortical vestibular evoked potential | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaswinder S Sandhu, Dr, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Trust, Sheffield, South Yorkshire, United Kingdom